CLINICAL TRIAL: NCT05717127
Title: Metabolic Impact of Intermittent Fasting in Early Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Caroline Kramer, Principal investigator, Endocrinologist and Clinician-scientist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-0299-A
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent fasting (time restricted feeding) (Experimental): Intermittent fasting (IF) study arm consisting of time restricted feeding with 20 hours of fasting and a 4 hour window of feeding (between 4 and 8 PM or between 5 to 9 PM).
  Interventions: Behavioral: Time restricted feeding
- Standard lifestyle (Active Comparator): Standard lifestyle recommendation as per the Diabetes Canada guidelines, where participants are encouraged to maintain regularity in timing and spacing of means with no specific recommendations regarding the hours of fasting
  Interventions: Behavioral: Standard lifestyle

INTERVENTIONS:
Behavioral: Time restricted feeding — Restricted feeding with 20 hours of fasting and a 4 hour window of feeding (between 4 and 8 PM or between 5 to 9 PM).
  Arms: Intermittent fasting (time restricted feeding)
Behavioral: Standard lifestyle — Standard lifestyle recommendations
  Arms: Standard lifestyle

SUMMARY:
One known cause of type 2 diabetes (T2DM) is beta-cell dysfunction, which refers to the inability of the beta-cells of the pancreas to produce enough insulin for the body's needs. Unfortunately, no anti-diabetic medication or lifestyle intervention has been shown to prevent the worsening of beta-cell function over time. Interestingly, however, intermittent fasting (IF) - where no food is consumed over a period of time - has been shown to promote weight loss and improve cardio-metabolic function. In individuals with T2DM, it is also been shown to improve glycemic control (i.e. reduce the sugar levels). While no research has studied whether IF can improve pancreatic beta-cell function, the positive metabolic effects suggest that it could provide some benefit. The current study will evaluate whether IF can improve pancreatic beta-cell function in individuals with early T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with type 2 diabetes mellitus diagnosed within preceding 10 years
* Age 20-70 years inclusive
* Body mass index ≥ 25 kg/m2
* Diabetes treatment consisting of lifestyle only, metformin or dipeptidyl peptidase-4 (DPP-4) inhibitor either as monotherapy or in combination
* HbA1c value of 5.5 - 9.0% inclusive

Exclusion Criteria:

* Current diabetes treatment with insulin, glucagon-like peptide-1 receptor agonists, sodium-glucose co-transporter 2 (SGLT-2) and/or sulfonylureas
* Involvements in any other clinical study on lifestyle intervention or requiring drug therapy
* Any history or eating disorder
* Renal dysfunction as evidenced by estimated glomerular filtration rate <45 mL/min by Modification of Diet in Renal Disease (MDRD) formula
* Hepatic disease considered to be clinically significant (includes jaundice, chronic hepatitis, or previous liver transplant) or transaminases >2.5x the upper limit of normal
* Malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy within the previous 5 years (with the exception of basal cell skin cancer)
* Any other factor likely to limit adherence to the study, in the opinion of the investigators

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Pancreatic beta-cell function | at week 16
  The difference in percentage change in beta-cell function between each intervention period, measured using the Insulin Secretion-Sensitivity Index-2 (ISSI-2)

SECONDARY OUTCOMES:
Fasting glucose | at week 16
  Difference in change in fasting glucose between each intervention period

OTHER OUTCOMES:
BMI | at week 16
  Difference in change in BMI between each intervention period
Waist circumference | at week 16
  Difference in change in waist circumference between each intervention period
Central abdominal fat mass on Dual X-ray Absorptiometry (DEXA) | at week 16
  Difference in change in central abdominal mass between each intervention period
Insulin sensitivity | at week 16
  Difference in insulin sensitivity measured by the Matsuda Index between each intervention period
Satiety | at week 16
  Difference in hunger assessed by Visual Analogue Scales (0 to 10mm with increased values associated with increased hunger) between each intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- Leadership Sinai Centre foe Diabetes - Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kramer CK, Zinman B, Feig DS, Retnakaran R. Effect of Time-Restricted Eating on beta-Cell Function in Adults With Type 2 Diabetes. J Clin Endocrinol Metab. 2025 May 19;110(6):e2045-e2053. doi: 10.1210/clinem/dgae594. PMID 39193706